CLINICAL TRIAL: NCT01842529
Title: Botulinum Toxin Injection in Epicardial Fat Pads Can Prevent Recurrences of Atrial Fibrillation After Cardiac Surgery: Randomized Pilot Study
Brief Title: Botulinum Toxin Injection in Epicardial Fat Pads To Treat Atrial Fibrillation After Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BT13-01
Record Dates: First submitted 2013-04-22; First posted 2013-04-29 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Paroxysmal Atrial Fibrillation; Indications for CABG
MeSH Terms: conditions — Atrial Fibrillation | interventions — Botulinum Toxins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CABG+ Botulinum toxin (Active Comparator): All patients underwent conventional CABG. After the main stage of the surgery botulinum toxin (Xeomin, incobotulinumtoxin A, Merz Pharma GmbH & Co KGaA, Germany; 50 U/1 mL at each fat pad; botulinum toxin group) was injected into the entire four visible area of the major epicardial fat pads. First epicardial left atrial fat pad is located anterior to the right superior pulmonary vein and corresponding to the anterior right GP; second epicardial fat pad is located inferoposterior to the right inferior pulmonary vein and corresponding to the inferior right GP; third fat pad is located anterior to the left superior PV and left inferior PV (between the PVs and LAA), corresponding to the Marshall tract GP and superior left GP; forth fat pad located inferiorly to the left inferior PV and extends posteriorly and corresponding to the inferior left GP.
  Interventions: Biological: botulinum toxin injection; Device: Implantable loop recorder
- Control (Active Comparator): All patients underwent conventional CABG. After the main stage of the surgery 0.9% normal saline (1 mL at each fat pad; placebo group) was injected into the entire four visible area of the major epicardial fat pads. First epicardial left atrial fat pad is located anterior to the right superior pulmonary vein and corresponding to the anterior right GP; second epicardial fat pad is located inferoposterior to the right inferior pulmonary vein and corresponding to the inferior right GP; third fat pad is located anterior to the left superior PV and left inferior PV (between the PVs and LAA), corresponding to the Marshall tract GP and superior left GP; forth fat pad located inferiorly to the left inferior PV and extends posteriorly and corresponding to the inferior left GP.
  Interventions: Biological: 0.9% normal saline injection; Device: Implantable loop recorder

INTERVENTIONS:
Biological: botulinum toxin injection
  Arms: CABG+ Botulinum toxin
Biological: 0.9% normal saline injection
  Arms: Control
Device: Implantable loop recorder

SUMMARY:
The aim of this prospective randomized double-blind study was to compare the efficacy and safety of Botulinum toxin injection in epicardial fat pads for preventing recurrences (in early postoperative period) of atrial tachyarrhythmia in patients with paroxysmal atrial fibrillation undergoing coronary artery bypass graft (CABG) surgery.

ELIGIBILITY:
Inclusion Criteria:

* PAF
* Indication for CABG according to the American College of Cardiology/American Heart Association (ACC/AHA) guidelines for CABG surgery

Exclusion Criteria:

* Previous heart surgery and AF ablation procedure
* Emergency CABG
* Unstable angina or heart failure
* Persistent AF, AF at the time of screening (planned Maze procedure or pulmonary vein isolation)
* Use of I or III antiarrhythmic drugs within 5 elimination half-lives of the drug (or within 2 months for amiodarone)
* Requiring concomitant valve surgery
* Left ventricle ejection fraction <35%
* Left atrial diameter >55 mm
* Unwillingness to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
recurrence of > 30 secs of atrial tachyarrhythmia, including AF and atrial flutter/tachycardia, after CABG procedure on no antiarrhythmic drug | 1 year

SECONDARY OUTCOMES:
time intervals from end of surgery to weaning from ventilation, extubation and discharge from ICU | 1 year
post-CABG length of stay | 12 months
incidence of congestive heart failure | 12 months
incidence of sustained ventricular arrhythmias | 12 months
incidence of myocardial infarction | 12 months
incidence of renal failure | 12 months
incidence of respiratory failure | 12 months
stroke or transient ischemic attack | 12 months
rehospitalization | 12 months
readmission to ICU | 12 months
number of deaths | 12 months
post-CABG length of stay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, FESC, Principal Investigator — State Research Institute of Circulation Pathology
Locations (3):
- The Valley Health System and Columbia University College of Physicians & Surgeons, New York, New York, United States
- Russia (2):
  - State Research Institute of Circulation Pathology, Novosibirsk
  - Institute of Cardiology, Siberian Division of Russian Academy of Medical Sciences, Tomsk

REFERENCES:
- [Derived] Romanov A, Pokushalov E, Ponomarev D, Bayramova S, Shabanov V, Losik D, Stenin I, Elesin D, Mikheenko I, Strelnikov A, Sergeevichev D, Kozlov B, Po SS, Steinberg JS. Long-term suppression of atrial fibrillation by botulinum toxin injection into epicardial fat pads in patients undergoing cardiac surgery: Three-year follow-up of a randomized study. Heart Rhythm. 2019 Feb;16(2):172-177. doi: 10.1016/j.hrthm.2018.08.019. Epub 2018 Nov 7. PMID 30414841
- [Derived] Pokushalov E, Kozlov B, Romanov A, Strelnikov A, Bayramova S, Sergeevichev D, Bogachev-Prokophiev A, Zheleznev S, Shipulin V, Lomivorotov VV, Karaskov A, Po SS, Steinberg JS. Long-Term Suppression of Atrial Fibrillation by Botulinum Toxin Injection Into Epicardial Fat Pads in Patients Undergoing Cardiac Surgery: One-Year Follow-Up of a Randomized Pilot Study. Circ Arrhythm Electrophysiol. 2015 Dec;8(6):1334-41. doi: 10.1161/CIRCEP.115.003199. Epub 2015 Oct 20. PMID 26486855
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru